CLINICAL TRIAL: NCT01664234
Title: Oxygen Insuflation and ArterialDesaturation During Tracheal Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Olga Plattner, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECS 1178/2012
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Infants; Difficult Airway
Keywords: infants with cleft palate; Pierre Robin; Treacher Collins; trisomy 21
MeSH Terms: conditions — Pierre Robin Syndrome; Mandibulofacial Dysostosis; Down Syndrome | interventions — Laryngoscopy; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- laryngoscopy with simultaneous insufflation of oxygen (Experimental): Patients will be randomly assigned to laryngoscopy with or without simultaneous insufflation of oxygen at 4 L/minute. Oxygen will be provided by a flowmeter connected via rigid tubing to the track-mounted endotracheal tube on the AirTraq.
  Interventions: Other: laryngoscopy with oxygen
- laryngoscopy without simultaneous oxygen insufflation (Placebo Comparator): Patients will be randomly assigned to laryngoscopy with or without simultaneous insufflation of oxygen at 4 L/minute. Oxygen will be provided by a flowmeter connected via rigid tubing to the track-mounted endotracheal tube on the AirTraq.
  Interventions: Other: laryngoscopy without oxygen

INTERVENTIONS:
Other: laryngoscopy with oxygen — Patients will be randomly assigned to laryngoscopy with or without simultaneous insufflation of oxygen at 4 L/minute. Oxygen will be provided by a flowmeter connected via rigid tubing to the track-mounted endotracheal tube on the AirTraq.
  Arms: laryngoscopy with simultaneous insufflation of oxygen
Other: laryngoscopy without oxygen — Patients will be randomly assigned to laryngoscopy without simultaneous insufflation of oxygen at 4 L/minute.
  Arms: laryngoscopy without simultaneous oxygen insufflation

SUMMARY:
Infants (0-1 yr.) with anticipated difficult airways will be enrolled in the study. Specifically, we will include infants with cleft palate, Pierre Robin, Treacher Collins, trisomy 21, or similar congenital malformations. Patients with American Society of Anesthesiologists physical status scores ≥3 will be excluded, as will those with congenital heart disease and left-to-right shunting. Patients will be randomly assigned to laryngoscopy with or without simultaneous insufflation of oxygen at 4 L/minute. Oxygen will be provided by a flowmeter connected via rigid tubing to the track-mounted endotracheal tube on the AirTraq. Randomization (1:1) will be based on computer-generated codes with random block sizes and stratified by hospital; allocation will be concealed and provided to clinicians via a secure web site that will be accessed shortly before induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* infants (0-2) difficult airways

Exclusion Criteria:

* . Patients with American Society of Anesthesiologists physical status scores ≥3 congenital heart disease left-to-right shunting

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
time to oxygen saturation | Day 1
  The randomized groups will be compared on time between laryngoscope (airtraq) insertion and reaching an oxygen saturation of 90%using a 2-tailed t-test or Wilcoxon-Mann-Whitney test, as appropriate.

SECONDARY OUTCOMES:
mean oxygenation comparison | Day 1
  Randomized groups will be compared on mean oxygen saturation at the time of intubation using a 2-sample t-test

CONTACTS AND LOCATIONS:
Overall Officials: Olga Plattner, M.D., Principal Investigator — Medizinischen Universität Wien Vienna
Locations (1):
- Medizinischen Universität Wien, Vienna, Borschkegasse, Austria